CLINICAL TRIAL: NCT01907490
Title: A Safety and Pharmacokinetic Study of Ha44 Gel Administered Topically Under Maximal Use Conditions for the Treatment of Head Lice Infestation.
Brief Title: Safety and PK Study of Ha44 Gel Under Maximal Use Conditions for Treatment of Head Lice Infestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Accelovance (Industry); Target Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ha03-004
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Head Lice Infestation
Keywords: Topical treatment of Head Lice Infestation
MeSH Terms: interventions — Benzyl Alcohol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Ha44 Gel 0.74%, topical solution, maximum feasible amount applied for 10 minutes
  Interventions: Drug: Ha44 Gel

INTERVENTIONS:
Drug: Ha44 Gel — Eligible subjects will be treated at the study site on Day 0 with a single application of the maximum feasible amount of Ha44 Gel, to ensure saturation of the scalp and hair.
  Other Names: Benzyl Alcohol

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a single application of Ha44 Gel 0.74% w/v for the treatment of head lice under maximal use conditions.

Secondary objective is to evaluate pharmacokinetics of Ha44 and benzyl alcohol (contained in Ha44 vehicle) under maximal use conditions.

DETAILED DESCRIPTION:
This is an open-label safety and pharmacokinetic (PK) study involving a single application of Ha44 Gel 0.74% administered under maximal use conditions.

All participants must have an active head lice infestation (at least 3 live lice) and be 6 months to 17 years of age. The study will enroll approximately 36 pediatric subjects between the ages of 6 months and 17 years.

Pediatric PK samples will be collected at 0 (predose), 30 and 60 mins and 2 and 8 hrs time points.

More than one household member with an active lice infestation may participate in the study. Eligible subjects will be consented and screened for study eligibility on Day 0 (Visit 1). All subjects will return to the study site for three follow-up clinic visits at Days 1, 7 and 14. The maximum study duration for a subject is 16 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 6 months to 17 years of age
3. Be in good health, as determined by medical history and physical examination
4. Has an active head lice infestation at screening as determined by an experienced evaluator. An active infestation is defined as the presence of at least 3 live lice.
5. Female subjects must be:

   * Of non-childbearing potential (no history of menstrual periods, post-hysterectomy, or post-menopausal for at least 2 years) OR,
   * If of childbearing potential, must have a negative urine pregnancy test prior to treatment and agree to use a highly effective method of contraception from Day 0 through the Day 14 visit. Acceptable methods of contraception include abstinence, vasectomized partner, tubal ligation, combined oral hormonal contraceptive, contraceptive injection, contraceptive patch, or IUD. If a hormonal contraception is the only method, the subject must have been on a stable dose for at least 3 months.
6. The parent/guardian agrees to allow serial blood samples collected from subject for PK analysis during study.
7. Has signed an informed consent and/or assent form (ICF).

Exclusion Criteria:

1. Has a condition or illness that, in the opinion of the Investigator, may interfere with the study results.
2. Has current dermatological disease or inflammation on the face, scalp, ears, neck or back, including eczema, atopic dermatitis, alopecia, psoriasis or any other chronic skin disease that, in the opinion of the Investigator, would interfere with the safety or PK evaluation.
3. Had a prior reaction to products containing piperonyl butoxide, pyrethrin, or pyrethrum extract.
4. Has been using hormonal contraception for less than 3 months.
5. Is pregnant or currently nursing.
6. Receiving systemic or topical medication, which in the opinion of the Investigator, may interfere with the study results.
7. Has received an investigational agent within 30 days prior to Day 0.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ha44 Gel 0.74% w/w: Ha44 Gel 0.74% w/w Open label, one arm
Period: Overall Study
Arm/Group | Ha44 Gel 0.74% w/w
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ha44 Gel 0.74% w/w
Number analyzed (Participants) | 38
Age, Customized [Number; unit: participants]
  6months-<12 months | 8
  12 months- <2 years | 9
  2 years - <3 years | 11
  3years-<18 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of the Subjects With AEs.
Description: Safety and tolerability assessed by AEs. Number of subjects with reporting AEs.
Time Frame: 3 months
Population: paediatric population, children between ages 6 months to <18 years.
Measure: Number; unit: participants
Arm/Group | Ha44 Gel 0.74% w/w
Number analyzed (Participants) | 38
participants | 8

2. Secondary Outcome: Pk Parameters: Cmax
Description: Maximum concentration of Ha44 (Cmax)
Time Frame: 0 to 8 hours
Population: Pharmacokinetic (PK) population included subjects who had sufficient concentration-time profiles for PK analyses.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- HA44 Gel 0.74%: Ha44 Gel 0.74%, topical solution, maximum feasible amount applied for 10 minutes
  Ha44 Gel: Eligible subjects were treated at the study site on Day 0 with a single application of the maximum feasible amount of Ha44 Gel, to ensure saturation of the scalp and hair.
Arm/Group | HA44 Gel 0.74%
Number analyzed (Participants) | 28
ng/mL | 141.4 [16 to 397]

3. Secondary Outcome: PK Parameters: Tmax
Description: Time to maximum concentration of Ha44 (Tmax)
Time Frame: 0-8 hours
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | HA44 Gel 0.74%
Number analyzed (Participants) | 28
hours | 0.8 [0 to 2]

4. Secondary Outcome: PK Parameters: AUC(0-8)
Description: Area under the concentration-time curve of Ha44 (AUC 0-8)
Time Frame: 0-8 hours
Population: PK Population
Measure: Mean (Full Range); unit: ng.h/mL
Arm/Group | HA44 Gel 0.74%
Number analyzed (Participants) | 28
ng.h/mL | 447.5 [80 to 971]

ADVERSE EVENTS:
Time Frame: From the time of IP application on Day 0 until Day 14
Description: Adverse events were systematically collected from the time of IP administration on Day 0 until Day 14.
Arm/Group | Ha44 Gel 0.74% w/w
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 2/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ha44 Gel 0.74% w/w (N=38)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For any publication or presentation the materials will be provided to the sponsor for approval. Sponsor will be permitted of 90-120 days for a review and shall have right to request modification if the material to be published will jeopardize the intellectual property of the sponsor .